CLINICAL TRIAL: NCT06042764
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of Novel Coronavirus Broad-spectrum Neutralizing Antibody SA55 Injection in the Treatment of Mild/Moderate COVID-19 Patients
Brief Title: SA55 Injection Phase II Study in the Treatment of Mild/Moderate COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-SA55-2001
Record Dates: First submitted 2023-08-26; First posted 2023-09-21 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Infection of Upper Respiratory Tract Caused by 2019-nCoV
Keywords: 2019-nCoV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SA55 Injection (Experimental): Group 1: 300 mg Group 2: 600 mg
  Interventions: Drug: SA55 Injection
- Placebo (Placebo Comparator): Group 1: 0 mg Group 2: 0 mg
  Interventions: Drug: SA55 Injection

INTERVENTIONS:
Drug: SA55 Injection — Novel coronavirus broad-spectrum neutralizing antibody SA55 injection (SA55 injection) is developed and produced by Beijing Kexing Zhongwei Biologics Technology Co., Ltd. The main component of SA55 injection is novel coronavirus broad-spectrum neutralizing antibody SA55. Each milliliter contains 150 mg of novel coronavirus broad-spectrum neutralizing antibody SA55. Excipients include histidine hydrochloride, arginine hydrochloride, histidine hydrochloride, sucrose, and polysorbate 80 (II)

SUMMARY:
Evaluating the efficacy and safety of SA55 injection in light/medium COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years on the day of enrollment;
* On the day of enrollment, novel coronavirus nucleic acid test was positive and/or novel coronavirus antigen test was positive;
* On the day of enrollment, it meets the criteria for mild or medium COVID-19 cases, and the time from the first COVID-19 infection related symptoms is within 72 hours;
* Within 24 hours before enrollment, one or more of the following symptoms or signs must be present: a. fever, b. cough, c. sore throat, d. nasal congestion/runny nose, e. headache, f. muscle pain, g. shortness of breath/difficulty breathing, h. nausea, i. fatigue, j. vomiting, k. diarrhea;
* Subjects (male and female of childbearing age) and their sexual partners voluntarily take effective contraceptive measures within 6 months after signing the informed consent form and administering the experimental drug, and do not have plans to donate sperm or eggs;
* At rest, when inhaling air, the oxygen saturation is greater than 93%;
* Subjects voluntarily participate in the experiment and sign an informed consent form before the start of the study.

Exclusion Criteria:

* Individuals who are known to be allergic to the investigational drug, any component in the preparation, or other similar drugs;
* Individuals weighing less than 40 kg;
* There are comorbidities that require surgery within one month, or comorbidities that are considered life-threatening within one month;
* Before screening, he has received neutralizing antibody drugs from COVID-19, or received human immunoglobulin or convalescent plasma treatment from convalescent patients within 3 months, or received small molecule drugs from COVID-19 within 7 days;
* Suspected or confirmed to have combined serious and active bacterial, fungal, viral or other infections (except for COVID-19 infection), such as acute systemic infection, the researcher believes that intervention measures may pose a risk;
* Individuals who tested positive for influenza A/B virus antigens during screening;
* Plan to become pregnant within 6 months, already pregnant, or breastfeeding;
* Participated in clinical trials of other drugs or medical devices within 3 months prior to screening;
* Having/having suffered from severe neurological disorders (epilepsy, convulsions, or seizures) or mental illness, or having a family history of mental illness;
* Suffering from/having previously suffered from severe neurological diseases or other serious illnesses that the researcher has determined to be unsuitable for participation in the study (including but not limited to current systemic infections, uncontrolled autoimmune diseases, uncontrolled immunodeficiency diseases, history of myocardial infarction or heart disease, etc.);
* Unable to cooperate with the follow-up of the study, or unable to guarantee the non use of concomitant drugs/vaccines/treatments prohibited by this protocol during the study period (see section 6.4.2);
* The researcher believes that due to other reasons, it is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of SA55 injection in mild or moderate COVID-19 patients | from baseline to D3, D5, D7
  Changes of novel coronavirus (SARS-CoV-2) load from baseline to D3, D5, D7

SECONDARY OUTCOMES:
Evaluate the safety of SA55 injection in mild or moderate COVID-19 patients | an average of 1 year
  The incidence of adverse events; The incidence of serious adverse events
Evaluation of the efficacy of SA55 injection in mild or moderate COVID-19 patients (impact on virological indicators) | (1) D9, D11, D15 (2) After administration (3) D3, D5, D7, D9, D11, D15
  (1) Changes in SARS-CoV-2 virus load relative to baseline at different time points; (2) Time to achieve continuous negative conversion of SARS-CoV-2 nucleic acid; (3) The proportion of subjects who achieved continuous negative SARS-CoV-2 nucleic acid conversion at different time points
Evaluation of the efficacy of SA55 injection in mild or moderate COVID-19 patients (impact on clinical indicators) | an average of 1 year
  Within 28 days after administration: the time of continuous disappearance of clinical symptoms and the time of continuous remission of clinical symptoms of 5, 7 and 11 COVID-19; The proportion of subjects who progress to severe/critically ill conditions; Hospitalization rate due to COVID-19; All cause mortality rate; Rescue treatment rate; Change of clinical symptom score of COVID-19 from baseline to different time points
Evaluate the pharmacokinetic characteristics of SA55 injection in mild or moderate COVID-19 patients | an average of 1 year
  Serum pharmacokinetic parameters of SA55 after medication (peak time Tmax, peak concentration Cmax, area under the drug time curve AUC0-t, AUC0- ∞, elimination half-life t1/2, apparent clearance rate CL/F, apparent distribution volume Vd/F, etc.)
Evaluation of serum COVID-19 neutralizing activity at different time points | an average of 1 year
  Serum pharmacokinetic parameters of SA55 after medication (peak time Tmax, peak concentration Cmax, area under the drug time curve AUC0-t, AUC0- ∞, elimination half-life t1/2, apparent clearance rate CL/F, apparent distribution volume Vd/F, etc.)
Evaluating the immunogenicity of SA55 injection | an average of 1 year
  Serum anti drug antibody (ADA) levels at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided